CLINICAL TRIAL: NCT00227032
Title: Phase I Study of Erlotinib Administered Every 72 Hours in Patients With Glioblastoma Multiforme With Pharmacokinetic/Pharmacodynamic Correlates
Brief Title: Erlotinib in Treating Patients With Progressive Glioblastoma Multiforme
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0424; CDR0000550155 (Other: PDQ number)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects receiving EIAEDs (Experimental): Patients will be stratified according to concurrent use of enzyme inducing anti-epileptic drugs (EIAED)
  Interventions: Drug: erlotinib hydrochloride
- Subjects NOT taking EIAEDs (Experimental): Patients will be stratified according to concurrent use of enzyme inducing anti-epileptic drugs (EIAED)
  Interventions: Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride — 300 mg, per day for subjects taking EIAEDs
  150 mg, per day for those NOT taking EIAEDs

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of erlotinib in treating patients with progressive glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of erlotinib hydrochloride when administered in escalating doses every 72 hours in patients with progressive glioblastoma multiforme.

Secondary

* Determine the relationship between plasma and cerebrospinal fluid (CSF) concentrations of erlotinib hydrochloride in these patients.
* Determine the relationship between plasma and CSF concentrations of erlotinib hydrochloride in patients not receiving concurrent enzyme-inducing antiepileptic drugs (EIAEDs) vs those receiving concurrent EIAEDs.
* Correlate CYP3A4 activity, as measured by midazolam hydrochloride clearance, with plasma clearance of erlotinib hydrochloride in these patients.
* Correlate CYP1A2 activity, as measured by the 4-hour paraxanthine (17X)/caffeine (137X) plasma ratio, with plasma clearance of erlotinib hydrochloride in these patients.
* Determine, preliminarily, objective response and disease progression in patients treated with erlotinib hydrochloride.
* Correlate the presence of EGFRvIII mutation with objective response and disease progression in patients treated with erlotinib hydrochloride.

OUTLINE: This is an open-label, dose-escalation study. Patients are stratified according to use of concurrent enzyme-inducing antiepileptic drugs (EIAEDs) (yes vs no).

Patients receive oral erlotinib hydrochloride once every 72 hours for 28 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses* of erlotinib hydrochloride until the maximum tolerated dose (MTD) is determined or preliminary results show no direct relationship between plasma and cerebrospinal fluid concentrations. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

NOTE: *Interim enrollment of patients is allowed; these patients receive the current approved dose of erlotinib hydrochloride.

Patients undergo blood sample collection periodically on day 13 for pharmacokinetic studies. The pharmacokinetic study comprises midazolam hydrochloride and caffeine clearance assessment and correlation of these assessments with CYP3A4 activity and CYP1A2 activity.

Paraffin-embedded and frozen tumor tissue is obtained from patients who underwent prior surgical resection for analysis of wild-type EGFR and EGFRvIII mutation by immunohistochemistry.

Quality of life is assessed at baseline and then at 1 month and 6 months.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme (or high-grade glioma that is behaving clinically and/or radiographically like glioblastoma multiforme)
* Progressed after first-line therapy (e.g., surgery, chemotherapy, or radiotherapy)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* ANC > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 8.5 g/dL
* ALT and AST < 2 times upper limit of normal (ULN)
* Alkaline phosphatase < 2 times ULN
* Bilirubin < 1.5 mg/dL
* Creatinine < 1.5 mg/dL OR creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No diagnosis or history of significant renal or hepatic disease
* No contraindication (e.g., mass effect, brain shift) to lumbar puncture procedure
* No active infection
* No diagnosis or history of corneal abnormalities
* No diagnosis or history of malabsorptive syndrome or other disorder affecting gastrointestinal absorption
* No history of hypersensitivity reactions to midazolam hydrochloride (CYP3A4 biomarker)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 12 months
  Progression -free survival will be measured by radographic response using RECIST critera.
Correlation between presence of the EGFRvIII mutation with treatment outcomes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Lindley, PharmD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Frances A. Collichio, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States